CLINICAL TRIAL: NCT07090720
Title: Melatonin Effects on the Left Ventricular Function in Neonates With Persistent Pulmonary Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Asmaa Mahmoud Abdel Hamid Elmesiry, Lecturer of Pediatrics, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36173//12/22
Record Dates: First submitted 2025-07-21; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Melatonin; Left Ventricular Function; Neonates; Persistent Pulmonary Hypertension
MeSH Terms: interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Experimental): Neonates were given Melatonin.
  Interventions: Drug: Melatonin
- Group II (Placebo Comparator): Neonates received placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Melatonin — Neonates were given Melatonin.
  Arms: Group I
Other: Placebo — Neonates received placebo.
  Arms: Group II

SUMMARY:
This study aimed to evaluate the effect of melatonin on the left ventricular function in neonates with persistent pulmonary hypertension

DETAILED DESCRIPTION:
Persistent pulmonary hypertension of the newborn (PPHN) is a potentially deadly disorder in which the circulation of the fetus is unable to adjust to the extrauterine environment. Persistently high pulmonary pressures may cause right-to-left shunting, hypoxia, and right ventricular failure.

Melatonin, a neurohormone produced by the pineal gland, offers an exceptional defense against reactive oxygen species (ROS). Infants are unable to synthesize melatonin during their first few weeks of life, which may exacerbate oxidative stress in hypoxic conditions. Additionally, Melatonin's antioxidative capabilities have been shown in neonatal pulmonary and respiratory disorders.

ELIGIBILITY:
Inclusion Criteria:

* Neonates of ≥ 36 weeks of gestational age.
* Both sexes.
* Admitted with persistent pulmonary hypertension.

Exclusion Criteria:

* Preterm infants < 36 weeks of gestation.
* Infants with congenital heart diseases.
* Infants with dysrhythmia.
* Chromosomal abnormalities.
* Severe pathological jaundice.
* Metabolic or endocrinal disorders.
* Major congenital malformations.

Min Age: 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Left ventricle global longitudinal strain | Immediately after medication (Up to 1 hour)
  Left ventricle global longitudinal strain (LV-GLS) was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.